CLINICAL TRIAL: NCT07311772
Title: A Randomized Controlled Study of Houyanqing Oral Liquid Combined With Conventional Treatment Versus Conventional Treatment Alone for Preventing and Treating Radiation-Induced Oral Mucositis in Nasopharyngeal Carcinoma
Brief Title: Prevention and Treatment of Radiation-Induced Oral Mucositis in NPC With Houyanqing Oral Liquid
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Collaborators: Fujian Cancer Hospital (Other Government); Eye & ENT Hospital of Fudan University (Other); Zhejiang Cancer Hospital (Other); West China Hospital (Other); Yunnan Cancer Hospital (Other); First Affiliated Hospital of Kunming Medical University (Other); The First People's Hospital of Changzhou (Other); Xiangya Hospital of Central South University (Other); Affiliated Cancer Hospital of Shantou University Medical College (Other); Wuzhou Red Cross Hospital (Other); Hunan Cancer Hospital (Other); Cancer Hospital of Guangxi Medical University (Other); Affiliated Cancer Hospital & Institute of Guangzhou Medical University (Other); Sun Yat-sen University Cancer Centre (Unknown); Cancer Hospital Chinese Academy of Medical Science (Unknown); The Fifth Affiliated Hospital, Sun Yat-sen University (Unknown)
Responsible Party: Principal Investigator, Ming-Yuan Chen, Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: ZDWY-CMY-Houyanqing OL
Record Dates: First submitted 2025-12-11; First posted 2025-12-31 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Nasopharyngeal Cancinoma (NPC); Radiation-induced Oral Mucositis
Keywords: Nasopharyngeal Cancinoma; Radiation-induced Oral Mucositis; Houyanqing Oral Liquid

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Houyanqing Oral Liquid combined with Conventional Treatment (Experimental): This arm involves Houyanqing Oral Liquid combined with conventional treatment for preventing radiation-induced oral mucositis (RIOM) in nasopharyngeal carcinoma patients receiving radical radiotherapy. Specific interventions include: 1) Houyanqing Oral Liquid administration before and during radiotherapy; 2) Conventional treatment (same as the control arm): oral hygiene management, epithelial repair promotion, and symptomatic support therapy; 3) Radical radiotherapy (conventional fractionation). The aim is to evaluate the effect of this combined regimen on reducing RIOM severity.
  Interventions: Drug: Houyanqing Oral Liquid; Other: Conventional Treatment for Radiation-Induced Oral Mucositis
- Conventional Treatment (Active Comparator): This arm consists of conventional treatment for preventing radiation-induced oral mucositis (RIOM) in nasopharyngeal carcinoma patients undergoing radical radiotherapy. Specific interventions include: 1) Oral hygiene management; 2) Epithelial repair promotion; 3) Symptomatic support . Patients in this arm will receive radical radiotherapy (conventional fractionation) but will not be administered Houyanqing Oral Liquid.
  Interventions: Other: Conventional Treatment for Radiation-Induced Oral Mucositis

INTERVENTIONS:
Drug: Houyanqing Oral Liquid — Houyanqing Oral Liquid is a Chinese herbal preparation formulated with Achyranthes aspera L., Kalimeris indica (L.) Sch.-Bip., Plantago asiatica L., and Carpesium abrotanoides L.. For this study, it is used in nasopharyngeal carcinoma patients receiving radical radiotherapy: the dosage is 10mL per administration, 4 times daily. The medication is initiated prior to radiotherapy and continued until the completion of radiotherapy, with the purpose of preventing and treating radiation-induced oral mucositis.
  Arms: Houyanqing Oral Liquid combined with Conventional Treatment
Other: Conventional Treatment for Radiation-Induced Oral Mucositis — This intervention refers to the conventional management measures for radiation-induced oral mucositis (RIOM) in nasopharyngeal carcinoma patients undergoing radical radiotherapy, including three modules: 1) Oral hygiene management; 2) Epithelial repair promotion; 3) Symptomatic support. These measures are implemented throughout the radiotherapy period to alleviate RIOM-related symptoms.

SUMMARY:
To explore the efficacy of Houyanqing Oral Liquid combined with conventional treatment in preventing and treating radiation-induced oral mucositis, so as to improve the quality of life of nasopharyngeal carcinoma patients received radiotherapy.

DETAILED DESCRIPTION:
Nasopharyngeal carcinoma (NPC) is a highly prevalent malignant tumor in China. Radical radiotherapy serves as its core treatment modality, yet radiation-induced oral mucositis (RIOM) is the most common adverse reaction of radiotherapy, with an incidence rate as high as 85%-100%, among which 34% of patients develop grade 3-4 mucositis. RIOM can cause oral pain, ulcers, and dysphagia, which not only severely reduce patients' quality of life but also may lead to radiotherapy interruption, increased infection risk, and elevated treatment costs. Therefore, the prevention and treatment of RIOM are of great significance.

At present, conventional clinical prevention and treatment methods include oral hygiene maintenance, epithelial repair-promoting drugs (e.g., recombinant human epidermal growth factor spray, sodium aescinate for injection), and symptomatic supportive care, but there is no universally recognized standard regimen. Houyanqing Oral Liquid is a traditional Chinese medicine preparation composed of Achyranthes aspera L., Kalimeris indica (L.) Sch.-Bip., Plantago asiatica L., and Carpesium abrotanoides L. It possesses the effects of clearing heat and detoxifying, relieving sore throat and pain. Previous studies have confirmed that it exhibits significant efficacy in anti-inflammation, bacteriostasis, and mucosal injury repair, which can shorten the course of oral ulcers and reduce the recurrence rate.

This study intends to conduct a randomized controlled clinical trial to compare the efficacy of Houyanqing Oral Liquid combined with conventional treatment versus conventional treatment alone in preventing RIOM in NPC patients. It aims to verify the advantages of the combined regimen in reducing the incidence of ≥ grade II RIOM, delaying the onset time, alleviating the severity of injury, and improving patients' quality of life, so as to provide a more effective and safe prevention and treatment strategy for RIOM in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

1. Staged as Stage I-IV according to the 9th edition of the TNM Classification of Malignant Tumors formulated by the American Joint Committee on Cancer (AJCC) and the Union for International Cancer Control (UICC);
2. Age: 18 to 75 years old;
3. Karnofsky Performance Status (KPS) score ≥ 80 before treatment;
4. No oral diseases (such as oral mucositis or salivary gland damage) before radiotherapy;
5. Requiring radical radiotherapy;
6. The patient has signed the informed consent form and is willing and able to comply with the study's follow-up visits, treatment plan, laboratory tests, and other research procedures.

Exclusion Criteria:

1. Patients with confirmed tumor recurrence, distant tumor metastasis, or who have received other anti-tumor treatments;
2. Previous history of head and neck radiotherapy;
3. Known allergy to the drugs used in this study (Houyanqing Oral Liquid, any conventional treatment drugs);
4. Local use of Houyanqing Oral Liquid, Recombinant Human Epidermal Growth Factor (rhEGF) Topical Solution, Vitamin B12 Solution, or Granulocyte-Macrophage Colony-Stimulating Factor (GM-CSF) mouthwash in the oral cavity within one month before enrollment;
5. Comorbidities requiring long-term treatment with immunosuppressive drugs, or systemic/local use of corticosteroids at immunosuppressive doses before enrollment;
6. HIV-positive patients;
7. Pregnant women or lactating women;
8. Patients with severe mental illnesses;
9. Patients with severe cardio-cerebrovascular diseases, endocrine disorders, infectious diseases, or other tumors.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 244 (Estimated)
Dates: Start 2025-12-15 (Estimated); Primary Completion 2027-03-15 (Estimated); Study Completion 2027-08-15 (Estimated)

PRIMARY OUTCOMES:
Incidence of ≥ Grade II radiation-induced oral mucositis | From the start of radical radiotherapy to the 3 months after the completion of radiotherapy
  The proportion of patients in the group who develop Grade II or above radiation-induced oral mucositis from the start of radiotherapy. The degree of oral mucosal damage is evaluated according to the Radiation Therapy Oncology Group/European Organization for Research and Treatment of Cancer (RTOG/EORTC) diagnostic and grading criteria for radiation-induced oral mucositis.

SECONDARY OUTCOMES:
Time to onset of Grade II or above radiation-induced oral mucositis | From the start of radical radiotherapy to the 3 months after the completion of radiotherapy.
  Time from the first day of radiotherapy to the first occurrence of Grade II or above radiation-induced oral mucositis according to RTOG/EORTC criteria.
Cumulative radiotherapy dose at onset of Grade II or above radiation-induced oral mucositis | From the start of radical radiotherapy to the 3 months after the completion of radiotherapy.
  Cumulative radiotherapy dose from the first day of radiotherapy to the first occurrence of Grade II or above radiation-induced oral mucositis according to RTOG/EORTC criteria.
Remission rate of Grade II or above radiation-induced oral mucositis | From the first occurrence of Grade II or above radiation-induced oral mucositis to 3 months after the completion of radiotherapy
  The proportion of patients who experience remission from Grade II or above to below Grade II radiation-induced oral mucositis after the first occurrence.
Complete remission rate of radiation-induced oral mucositis | From the first occurrence of Grade II or above radiation-induced oral mucositis to 3 months after the completion of radiotherapy
  The proportion of patients who achieve complete remission of Grade II or above radiation-induced oral mucositis after the first occurrence.
Remission time of Grade II or above radiation-induced oral mucositis | From the first occurrence of Grade II or above radiation-induced oral mucositis to 3 months after the completion of radiotherapy.
  Time from the first occurrence of Grade II or above radiation-induced oral mucositis to remission below Grade II.
Complete remission time of radiation-induced oral mucositis | From the first occurrence of Grade II or above radiation-induced oral mucositis to 3 months after the completion of radiotherapy.
  Time from the first occurrence of Grade II or above radiation-induced oral mucositis to complete remission.

CONTACTS AND LOCATIONS:
Overall Officials: Ming-Yuan Chen, MD, PhD, Principal Investigator — Fifth Affiliated Hospital of Sun Yat-sen University
Locations (16):
- China (16):
  - Cancer Hospital Chinese Academy of Medical Science, Beijing, Beijing Municipality
  - Fujian Medical University Cancer Hospital, Fuzhou, Fujian
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - Affiliated Cancer Hospital & Institute of Guangzhou Medical University, Guangzhou, Guangdong
  - Cancer Hospital of Shantou University Medical College, Shantou, Guangdong
  - Fifth Affiliated Hospital of Sun Yat-sen University, Zhuhai, Guangdong
  - Cancer Hospital of Guangxi Medical University, Nanning, Guangxi
  - Wuzhou Red Cross Hospital, Wuzhou, Guangxi
  - Xiangya Hospital of Central South University, Changsha, Hunan
  - Hunan Cancer Hospital, Changsha, Hunan
  - The First People's Hospital of Changzhou, Changzhou, Jiangsu
  - Eye & ENT Hospital of Fudan University, Shanghai, Shanghai Municipality
  - West China Hospital of Sichuan University, Chengdu, Sichuan
  - The First Affiliated Hospital of Kunming Medical University, Kunming, Yunnan
  - Yunnan Cancer Hospital, Kunming, Yunnan
  - Zhejiang Cancer Hospital, Hangzhou, Zhengjiang

IPD SHARING:
Plan to Share IPD: Undecided